CLINICAL TRIAL: NCT06987188
Title: Effects of Modified Pilates on Improving Trunk Control and Balance in Children With Mild Intellectual Disability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/24/0758
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Mild Intellectual Disability
Keywords: Mild Intellectual Disability; Trunk control; Balance; Physical therapy; pilate exercises

STUDY DESIGN:
Intervention Model Description: This study will be randomized controlled trial, conducted in Mind spark clinic, Lahore. This study will be completed in time duration of 8 weeks after the approval of synopsis. Non-probability convenience sampling technique will be used and 40 participants will be recruited in this study. Participants will be divided into two groups. Group A (Modified Pilates Exercises) and Group B (General Physiotherapy Plan). Tools will be used are Trunk control measurement (TCMS) and Pediatric Balance Scale (PBS). The data will be recorded at the baseline and after 8th week of intervention. After collection, data will be analyzed by using SPSS version 25.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): : Modified Pilates Exercises, will be given for 8 weeks, 4 times per week. Diaphragmatic Breathing, Bridging and Planks will be given. Intervention Session will be 40-45 minutes with short resting intervals
  Interventions: Other: Modified Pilate Exercises; Other: General Physiotherapy Plan
- Group B (Experimental): General Physiotherapy plan, Will be given for 8 weeks, 4 times per week. Bottom up Exercises, Bridging and Turning over facilitation. Intervention Session will be 40-45 minutes with short resting intervals
  Interventions: Other: Modified Pilate Exercises; Other: General Physiotherapy Plan

INTERVENTIONS:
Other: Modified Pilate Exercises — Modified Pilates exercises are gentle adaptations of traditional Pilates movements, designed to accommodate various fitness levels, physical limitations, or specific health conditions. These exercises focus on core strength, flexibility, posture, and controlled breathing while reducing strain on joints and muscles. Often recommended for beginners, seniors, or individuals recovering from injury or surgery, modified Pilates may involve the use of props like pillows, resistance bands, or chairs to support proper alignment and ease of movement. By emphasizing slow, mindful motions and personalized adjustments, modified Pilates helps individuals safely build strength, improve mobility, and enhance overall body awareness without the risk of overexertion.
Other: General Physiotherapy Plan — A general physiotherapy plan for improving trunk control and balance focuses on enhancing core stability, postural alignment, and coordinated movement through targeted exercises and functional activities. The plan typically begins with gentle activation of deep core muscles such as the transverse abdominis and pelvic floor, progressing to dynamic tasks that challenge balance and coordination, like seated weight shifts, bridging, and reaching tasks in various positions (sitting, kneeling, or standing). Balance training may include exercises on unstable surfaces, gait training, and proprioceptive activities to improve body awareness and stability. The physiotherapy approach is individualized, gradually increasing in complexity and intensity as the patient gains strength and confidence, with consistent emphasis on proper technique, breathing, and safety to support overall mobility and independence.

SUMMARY:
This randomized controlled trial will be conducted at Spectrum Clinic, Lahore, over a duration of 8 weeks to assess the impact of Modified Pilates Exercises on trunk control in children with Intellectual Disability (ID). ID is characterized by below-average IQ and delays in cognitive and functional development, affecting independence and motor skills. Trunk control plays a crucial role in posture, movement coordination, balance, and daily activities. A total of 40 participants will be selected through non-probability convenience sampling and randomly assigned to two groups: Group A (Modified Pilates Exercises) and Group B (General Physiotherapy Plan). Outcomes will be measured using the Trunk Control Measurement Scale (TCMS) and Pediatric Balance Scale (PBS) at baseline and after 8 weeks. Data will be analyzed using SPSS version 25.

DETAILED DESCRIPTION:
Intellectual Disability (ID) is a condition in which individuals experience below-average IQ. Although a variety of terms, including learning disabilities and mental retardation have been used when referring to people who have impairments that impact on their cognitive and adaptive functioning. ID refers to the onset of delayed developmental milestones, which impact on intellectual and functional development, hence independent functioning is likely to be significantly lower than that of the average person during their lifetime. Trunk control can help children with intellectual disabilities meet developmental milestones by helping them to maintain posture, navigate their surroundings, coordinate body part movement, module fine motor control, initiate vestibule oculomotor reflexes, use their hands for various activities, remain seated without falling over and kept their body aligned while walking, running and jumping.

This study will be randomized controlled trial, conducted in Spectrum clinic, Lahore. This study will be completed in time duration of 8 weeks after the approval of synopsis. Non-probability convenience sampling technique will be used and 40 participants will be recruited in this study. Participants will be divided into two groups. Group A (Modified Pilates Exercises) and Group B (General Physiotherapy Plan). Tools will be used are Trunk control measurement (TCMS) and Pediatric Balance Scale (PBS). The data will be recorded at the baseline and after 8th week of intervention. After collection, data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years.
* Diagnosed with mild intellectual disability (IQ 50-70)
* Ability to follow instruction and participate in Pilates Exercises
* No significant physical or neurological conditions that could affect participants

Exclusion Criteria:

* Severe intellectual disability(IQ<50)
* Significant physical and neurological conditions (Cerebral palsy, Spinal Cord Injury)
* Visual and Hearing impairments that could impact participation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | Baseline, 4th week, 8th week
  The Trunk Control Measurement Scale (TCMS) is a standardized assessment tool used to measure trunk control in individuals with developmental delay, neurological disorders, or motor impairments. It evaluates posture maintenance, trunk stabilization, and movement across six subtasks, each rated on a scale from 0 to 4 or 0 to 5. The total score ranges from 0 to 24, offering a comprehensive evaluation of trunk control ability. The TCMS identifies specific areas of difficulty, tracks progress over time, and directs targeted interventions to enhance trunk control. Administration involves verbal instructions, visual demonstration, or physical guidance from the evaluator, with the participant performing each task up to three times, scored based on the best attempt
Pediatric Berg Balance Measurement Scale (PBBMS) | Baseline, 4th week, 8th week
  The Pediatric Berg Balance Measurement (PBBM) is a well-established tool used to assess balance and postural control in children aged 5-15 years. Developed by Berg and colleagues, it comprises 14 items that evaluate standing, sitting, and transitional movements. Scores on the PBBM range from 0 to 56, with higher scores indicating better balance abilities(20). This assessment typically takes 15-20 minutes to administer and is highly reliable and valid. Physiotherapists, occupational therapists, and researchers utilize the PBBM to evaluate balance impairments in children with developmental delays, injuries, or neurological conditions, and to track progress and intervention outcomes effectively.

CONTACTS AND LOCATIONS:
Overall Officials: Khansa Khizar, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Pinjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balayi E, Sedaghati P, Ahmadabadi S. Effects of neuromuscular training on postural control of children with intellectual disability and developmental coordination disorders : Neuromuscular training and postural control. BMC Musculoskelet Disord. 2022 Jul 2;23(1):631. doi: 10.1186/s12891-022-05569-2. PMID 35780104